CLINICAL TRIAL: NCT07033637
Title: Promoting Health Through Symbiosis: Exploring the Relationship Between Gut Microbiota, Probiotics, and Physical Activity in Older Adults
Brief Title: Probiotics and Active Aging: Enhancing Gut Health
Acronym: PAAEGH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jose Luis Felipe (Other)
Responsible Party: Sponsor-Investigator, Jose Luis Felipe, Senior Lecturer, University of Castilla-La Mancha
Organization: University of Castilla-La Mancha (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: IGOID3
Record Dates: First submitted 2025-06-05; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Gut -Microbiota; Older People; Physical Activity; Physical Fitness; Mental Health; Probiotic; Healthy
Keywords: older people; gut microbiota; physical activity
MeSH Terms: conditions — Motor Activity; Psychological Well-Being | interventions — Dietary Supplements

STUDY DESIGN:
Intervention Model Description: This interventional study follows a parallel assignment model with three distinct groups of older adults (≥60 years), each comprising 30 participants:
  Group 1 (Intervention Group): Participants engage in a structured physical activity program and later receive a probiotic supplement (AB-DR7).
  Group 2 (Control Group A): Sedentary participants who receive the probiotic supplement without engaging in physical activity.
  Group 3 (Control Group B): Sedentary participants who receive a placebo and do not engage in physical activity.
  The study is conducted over 18 weeks, divided into two main phases:
  First 12 weeks: Group 1 performs physical activity; Groups 2 and 3 maintain their usual sedentary lifestyle.
  Following 6 weeks: Groups 1 and 2 begin probiotic intake; Group 3 continues with placebo.
  The model is designed to evaluate the independent and combined effects of physical activity and probiotic supplementation on gut microbiota composition, physical condition, and quality of life in old
Who Masked: Participant, Outcomes Assessor
Masking Description: In this double-blind study, both participants and outcomes assessors are masked to the intervention assignment. The probiotic and placebo capsules are identical in appearance, taste, and packaging, ensuring that participants cannot distinguish between them. Outcomes assessors responsible for evaluating physical condition, microbiota composition, and quality of life are also blinded to group allocation to minimize assessment bias. The investigators administering the interventions are not blinded due to logistical requirements in distributing the correct supplement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention Group - Physical Activity + Probiotics (Experimental): Participants in this arm will engage in a structured physical activity program for 12 weeks, followed by a 6-week period during which they will continue the exercise regimen and begin daily intake of a probiotic supplement (AB-DR7, containing Lactiplantibacillus plantarum CECT 7481). The goal is to assess the combined effects of physical activity and probiotics on gut microbiota, physical condition, and quality of life in older adults.
  Interventions: Other: Dietary Supplement; Behavioral: Structured Physical Activity Program
- Control Group A - Sedentary + Probiotics (Active Comparator): Participants in this arm will maintain their usual sedentary lifestyle throughout the study. After the initial 12-week observation period, they will begin a 6-week daily intake of the same probiotic supplement (AB-DR7). This arm is used to evaluate the effects of probiotics alone on gut microbiota and health indicators in the absence of physical activity.
  Interventions: Other: Dietary Supplement
- Control Group B - Sedentary + Placebo (Placebo Comparator): Participants in this arm will maintain a sedentary lifestyle and receive a placebo capsule identical in appearance to the probiotic, but containing maltodextrin instead of Lactiplantibacillus plantarum. This group serves as the baseline comparator to assess the natural variation in outcomes without intervention.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Dietary Supplement — A daily oral capsule containing 1 x 10⁹ CFU of Lactiplantibacillus plantarum CECT 7481 (32.5 mg), microcrystalline cellulose (304.1 mg), and magnesium stearate (3.4 mg). Administered once daily before the main meal for 6 weeks. Used to evaluate its effects on gut microbiota and physical health in older adults.
  Arms: Control Group A - Sedentary + Probiotics; Intervention Group - Physical Activity + Probiotics
Other: Placebo — A daily oral capsule identical in appearance to the probiotic capsule, containing maltodextrin instead of Lactiplantibacillus plantarum. Administered once daily before the main meal for 6 weeks. Used to control for placebo effects in the assessment of probiotic efficacy.
  Arms: Control Group B - Sedentary + Placebo
Behavioral: Structured Physical Activity Program — A 12-week supervised physical activity program conducted at municipal sports centers. Participants engage in moderate-intensity exercise at least 2 times per week. Designed to assess the impact of physical activity on gut microbiota, physical condition, and quality of life in older adults.
  Arms: Intervention Group - Physical Activity + Probiotics

SUMMARY:
The general objective of this clinical trial is to assess the physical fitness and gut microbiota of older adults, thereby highlighting the importance of focusing on health maintenance. By making use of available resources and fostering collaboration among the elements involved in the study, more specific objectives can be defined:

1. To determine the state of the gut flora in older adults through the analysis of the intestinal microbiota.
2. To identify changes in the intestinal microbiota resulting from the intake of probiotics in older adults.
3. To evaluate the effects of the intestinal microbiota in older adults participating in a training programme.
4. To assess the physical fitness and perceived quality of life in older adults who engage in sport activities supported by technology.

Participants will:

* Perform physical tests such as the 6-Minute Walk Test (6MWT), the Timed Up and Go (TUG), and the Sit-to-Stand test.
* Complete wellbeing questionnaires to assess their perceived quality of life and health status.
* Complete dietary habit questionnaires.
* Provide stool samples for microbiota analysis.
* Take part in exercise interventions or placebo exercise sessions, depending on their assigned group.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 60 years or older.
* Residents of Castilla-La Mancha or Madrid.
* Able to provide informed consent.
* For the intervention group: enrolled in a municipal physical activity program with a minimum frequency of 2 sessions per week.
* Willing to participate in all assessments and follow study instructions.
* Consent: Participants must provide written informed consent to participate in the study.

Exclusion Criteria:

* Recent serious musculoskeletal injuries (e.g., muscle tears, ligament ruptures, fractures).
* Current symptoms during exercise such as chest pain, dizziness, or joint pain.
* Uncontrolled hypertension (≥160/100 mmHg).
* Recent cardiac failure or infectious disease (e.g., meningitis, hepatitis, flu).
* Chronic gastrointestinal diseases (e.g., Crohn's disease, ulcerative colitis, IBS).
* Regular use of medications affecting gut motility or microbiota (e.g., laxatives >3 times/week).
* Immunodeficiency (e.g., HIV, active cancer).
* Use of antibiotics (oral or parenteral) within 4 weeks prior to the study.
* Regular intake of probiotic supplements or foods (e.g., Actimel) within 2 weeks prior to the study.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in gut microbiota composition | Baseline, Week 12, Week 18
  Assessment of gut microbiota diversity and composition using 16S rRNA sequencing of stool samples. Alpha and beta diversity indices will be calculated to evaluate changes over time and between groups.

SECONDARY OUTCOMES:
Change in quality of life scores | Baseline, Week 12, Week 18
  The Short Form Health Survey - 12 items (SF-12) is a validated, self-reported instrument used to assess health-related quality of life. It generates two composite scores:
  * Physical Component Summary (PCS-12)
  * Mental Component Summary (MCS-12)
  Score range: Norm-based scoring with a mean of 50 and a standard deviation of 10 in the general population.
  Interpretation:
  * Scores above 50 indicate better-than-average health-related quality of life.
  * Scores below 50 indicate worse-than-average health-related quality of life
Change in gastrointestinal symptom scores | Baseline, Week 12, Week 18
  Measured using the GSRS (Gastrointestinal Symptom Rating Scale), which includes 15 items grouped into five symptom clusters.
  Score range: 1 to 7 Interpretation: Higher scores reflect greater severity of gastrointestinal symptoms.
Change in 6-minute walk test distance | Baseline, Week 12, Week 18
  Distance walked in meters during the 6-minute walk test to assess cardiorespiratory fitness.
  Unit of measure: meters
Change in handgrip strength | Baseline, Week 12, Week 18
  Measured using a hand dynamometer to assess upper body strength.
  Unit of measure: kilograms
Change in body fat percentage | Baseline, Week 12, Week 18
  Measured using bioimpedance analysis to assess body composition.
  Unit of measure: percent (%)
Change in balance performance | Baseline, Week 12, Week 18
  Measured using a pressure platform during a 30-second Romberg test. The outcome includes center of pressure displacement and bilateral weight distribution to assess balance and fall risk.
  Unit of measure: Sway Index

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to privacy concerns and the nature of the study being part of a doctoral thesis. The data are collected under strict confidentiality agreements and are intended solely for internal analysis and academic purposes within the research team. Any future data sharing would require additional ethical approvals and participant consent.

REFERENCES:
- [Background] Thomas E, Battaglia G, Patti A, Brusa J, Leonardi V, Palma A, Bellafiore M. Physical activity programs for balance and fall prevention in elderly: A systematic review. Medicine (Baltimore). 2019 Jul;98(27):e16218. doi: 10.1097/MD.0000000000016218. PMID 31277132
- [Background] Nascimento V, Fonseca C, Pinho LG, Lopes MJ. Person-Centered Health Intervention Programs, Provided at Home to Older Adults with Multimorbidity and Their Caregivers: Protocol for a Systematic Review. J Pers Med. 2022 Dec 23;13(1):27. doi: 10.3390/jpm13010027. PMID 36675688
- [Background] Marttinen M, Ala-Jaakkola R, Laitila A, Lehtinen MJ. Gut Microbiota, Probiotics and Physical Performance in Athletes and Physically Active Individuals. Nutrients. 2020 Sep 25;12(10):2936. doi: 10.3390/nu12102936. PMID 32992765
- [Background] Barnett K, Mercer SW, Norbury M, Watt G, Wyke S, Guthrie B. Epidemiology of multimorbidity and implications for health care, research, and medical education: a cross-sectional study. Lancet. 2012 Jul 7;380(9836):37-43. doi: 10.1016/S0140-6736(12)60240-2. Epub 2012 May 10. PMID 22579043
- [Background] Aya V, Jimenez P, Munoz E, Ramirez JD. Effects of exercise and physical activity on gut microbiota composition and function in older adults: a systematic review. BMC Geriatr. 2023 Jun 12;23(1):364. doi: 10.1186/s12877-023-04066-y. PMID 37308839